CLINICAL TRIAL: NCT00732966
Title: Ocsaar and CYP2C9 Ploymorphism, Is There a Connection Between Pharmacokinetics, Pharmacodynamics and Pharmacogenetics?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Koren Peleg Ronit MD, Assaf-Harofeh Medical Center internal medicine A
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ronit3
Record Dates: First submitted 2008-08-10; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension
Keywords: cyp2c9; losartan; pharmacogenetics; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Hypertension | interventions — Losartan; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hypertensive patients will be treated with losartan for one months
  Interventions: Drug: losartan; Drug: valsartan
- 2 (Experimental): Hypertensive patients will be treated with valsartan
  Interventions: Drug: losartan; Drug: valsartan

INTERVENTIONS:
Drug: losartan — with losartan 50 mg once daily for one month
Drug: valsartan — valsartan 160 mg once daily

SUMMARY:
Most Angiotensin receptor blocker's (ARBs) are metabolized by cytochrome P4502C9 (CYP2C9), one of the major isoforms of the cytochrome P450 in human liver microsome. The purpose of this study is to evaluate whether CYP2C9 polymorphism has a significant clinical influence on the blood pressure lowering effect of losartan and valsartan. Weather there is a genetic importance in choosing the right ARB for the right patient.

DETAILED DESCRIPTION:
Losartan, the first angiotentsin II receptor blocker (ARB), is known to reduce blood pressure (BP). The LIFE study, Cardiovascular Morbidity and Mortality in the Losartan Intervention for Endpoint Reduction, showed that losartan prevented more cardiovascular morbidity and mortality than the ß receptor blocker atenolol. This effect was independent of its BP lowering effect. Left ventricular hypertrophy (LVH) is known to be a cardinal manifestation of BP and an independent risk factor for cardiovascular complications. In the patient subgroup of isolated systolic hypertension, losartan was found to reduce cardiovascular and all cause mortality and to reverse LVH.

ARBs are used for the treatment of hypertension, alone or in combination with other antihypertensive drugs, such as calcium channel blockers, diuretics or angiotensin I converting enzyme (ACE) inhibitors. ACE inhibitors and ARBs may also have an important role in the prevention of type II diabetes and should be considered first line agents in hypertensive patients with impaired fasting glucose or metabolic syndrome.

Most ARBs are metabolized by cytochrome P4502C9 (CYP2C9), one of the major isoforms of the cytochrome P450 in human liver microsome. It converts losartan to its pharmacologically active metabolite EXP-3174 (E-3174). Other ARBs such as telmisartan and olmesartan are innate to CYP2C9, whereas candesartan and valsartan are metabolized by it to pharmacologically inactive metabolites. Maximal concentration of the drug is reached two hours post administration. Fourteen percent of the orally administered medication is converted to E-3174, which is 10 to 40 fold more potent than losartan. The pharmacokinetics of losartan and E-3174 are linear, dose dependent and do not change after repetitive administration. The CYP2C9 gene has three main polymorphic variations caused by single nucleotide polymorphism; the most common allele is CYP2C9*1 (Arg144 Ile359), and the two less common CYP2C9*2 (Cys 144Ile359) and CYP2CP*3 (Arg144Leu359) that code for an enzyme with decreased activity. The oxidation of losartan is decreased 2,3 and 40 fold in individuals genotyped as CYP2C9*1*3, CYP2C9*2*3 and CYP2C9*3*3 compared to individuals genotyped as CYP2C9*1*1.CYP2C9*3 was found to influence losartan's metabolism more than does CYP2C9*2.

The distribution of CYP2C9 allelic variants within different ethnic groups varies. In Caucasians the allele frequencies of CYP2C9*1, CYP2C9*2 and CYP2C9*3 have been reported to be 0.79-0.86, 0.08-0.135 and 0.03-0.085 respectively, whereas very low frequency of the alleles CYP2C9*2 and CYP2C9*3 have been reported in Asian populations (0 and 0.02-0.05 respectively). Ashkenazi Jews were found to have similar prevalence of allele polymorphism as North American Caucasian population (the CYP2C9*1, *2, *3 allele frequencies were 0.772, 0.140 and 0.086, respectively). Nakai K et al. evaluated the population prevalence of the different alleles in four different ethnic groups in the Israeli population: Ashkenazi, Moroccan, Libyan and Yemenite Jews. They found that in the Ashkenazi population, the prevalence of CYP2C9*1, CYP2C9*2 and CYP2C9*3 variants was 0.83, 0.17 and 0.15 respectively, in the Yemenite population 0.89, 0.1 and 0.15 respectively, in the Moroccan population 0.81, 0.19 and 0.23 respectively and in the Libyan population 0.69, 0.27 and 0.31 respectively.

Many drugs have been found to be substrates for CYP2C9, including fluoxetine, losartan, phenytoin, tolbutamide, torsemide, warfarin, and numerous NSAIDs. CYP2C9 activity is inducible by rifampicin and possibly also by carbamazepine, ethanol and phenobarbitone. Several drugs have been reported to inhibit CYP2C9 activity in vivo or in vitro, for example: fluconazole, amiodarone, trimethoprim, fluvastatin, cimetidine and chloramphenicol.

An in vitro study demonstrated that the clearance of losartan was reduced significantly in human liver microsomes obtained from CYP2C9*3*3 and CYP2C9*2*2 homozygous individuals, and from CYP2C9*3*1 heterozygous individuals but not from CYP2C9*2*1 individuals. In this study, no clear conclusion could be made regarding the CYP2C9*2*3 genotype. In another study, no influence of the CYP2C9 polymorphism on the pharmacokinetics of losartan or E-3174 was found after a single oral dose of 50 mg losartan.

Irbesartan undergoes metabolism through the CYP2C9 to an inactive metabolite. Hallberg P et al. randomly assigned 115 hypertensive patients to be treated with atenolol or irbesartan. They found that the CYP2C9 genotype predicted the BP response to irbesartan and had no influence on the effect of atenolol.

Purpose:

The purpose of this study is to evaluate whether CYP2C9 polymorphism has a significant clinical influence on the BP lowering effect of losartan and valsartan. Weather there is a genetic importance in choosing the right ARB for the right patient.

Methods

Patients:

A screening period will be conducted in which hypertensive patients aged 18 years and over, will undergo a genetic evaluation for CYP2C9 polymorphism.

Patients will sign a written informed consent before their inclusion in the study. No other change in patients' medication regimen will be made.

Study design:

The study will be a prospective non randomized trial. All patients fulfilling the inclusion and exclusion criteria will be treated with losartan 50 mg once daily for one month. After a wash out period of one week losartan treatment will be replaced with valsartan 160 mg once daily. Patients will be evaluated at baseline and following losartan and valsartan treatment. Patients will undergo a 24 hour ambulatory BP monitoring at baseline, one months following losartan treatment and one month following valsartan treatment. Creatinine and Potassium levels will be measeured at baseline and one week following each drug administration, blood sample will be collected to measure the losartan/ E-3174 ration.

Genetic evaluation:

Polymerase chain reaction amplification will be preformed with the use of specific primers. Genotyping of the polymorphic CYP2C9 genes will be made using real time PCR (RT PCR) technology with Roche light cycler. The procedure is made in a closed system which decreases the chance for contamination.

Losartan and E-3174 Analysis:

The losartan and e-3174 assays will be performed using a reversed phase high performance liquid chromatography (HPLC) method. Hewlett Packard HP-1090 Series II will be used.

ELIGIBILITY:
Inclusion Criteria:

* The study will include 30 patients with the 3 most prevalent alleles of CYP2C9 *1, *2 and*3, 10 patients of each group.

Exclusion Criteria:

* Patients treated with losartan or valsartan prior to their enrollment to the study,
* Patients with BP below 140 systolic or 90 diastolic in an ambulatory 24 hours BP monitoring, acute coronary syndrome during the 6 months previous to the study,
* Renal failure with creatinin levels above 1.5 mg/dL, hyperkalemia (K > 5 mg/dL),
* Hematologic or solid malignancies or pregnancy.
* Patients will also be excluded from the study if they are known to use one of the drugs inducing or inhibiting the CYP2C9, such as

  * rifampicin carbamazepine,
  * ethanol,
  * phenobarbitone,
  * fluconazole,
  * amiodarone,
  * trimethoprim,
  * fluvastatin,
  * cimetidine
  * chloramphenicol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Blood pressure lowering effect of losartan and valsartan in patients with different CYP2C9 allels | one month

SECONDARY OUTCOMES:
losartan/E-3174 ratio in different allelic groups of CYP2C9 | one month

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Koren Peleg, MD, Principal Investigator — Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine, Tel Aviv, Israel